CLINICAL TRIAL: NCT05367453
Title: Nutritional Clinical Trial to Evaluate the Regular Consumption Effect of a Probiotic With High Beta-galactosidase Activity Over Lactose Intolerance Gastrointestinal Symptoms in Patients With Lactose Intolerance
Brief Title: Effect of a Probiotic With High Beta-galactosidase Activity on Patients With Lactose Intolerance
Acronym: PROBIOLAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Go Fruselva, S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HULP 5758
Record Dates: First submitted 2022-04-18; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-02

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance | interventions — Probiotics; Lactase; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactase (Active Comparator): Volunteers will consume once a day for 1 month a tropical juice (orange, mango, pineapple and turmeric) and a lactase tablet
  Interventions: Other: a Tropical juice with no probiotics; Other: lactase tablet
- Probiotic (Experimental): Volunteers will consume once a day for 1 month the probiotic added to a liquid matrix (tropical juice) and and a placebo tablet (cornstarch)
  Interventions: Dietary Supplement: Tropical juice with probiotics (B.coagulans); Other: placebo tablet (cornstarch)

INTERVENTIONS:
Dietary Supplement: Tropical juice with probiotics (B.coagulans) — Once a day during all the intervention phase, volunteers with lactose intolerance should allow the spore-forming ability of B. coagulans in order to digest lactase from dairy products through regular consumption of Tropical juice with probiotics (B.coagulans)
  Arms: Probiotic
Other: a Tropical juice with no probiotics — Once a day during all the intervention phase, volunteers with lactose intolerance should consume a Tropical juice with no probiotics
  Arms: Lactase
Other: lactase tablet — lactase tablet
  Arms: Lactase
Other: placebo tablet (cornstarch) — placebo tablet (cornstarch)
  Arms: Probiotic

SUMMARY:
Lactose intolerance is a chronic disease caused by the total/partial lack of lactase production. When lactose is not properly digest, it is consumed by the microbiota. This situation presents different gastrointestinal symptoms such as meteorism, pain, bloating, diarrhoea and nausea. The dietetic treatment for this patients consists of avoiding lactose-rich foods, mainly milk and dairy products. However, nowadays exists a large diversity of lactose-free products specially focused on lactose intolerants. In this context, using B.coagulans as a probiotic in a food matrix could be an alternative for these patients, since its ability of spore forming and the production of beta-galactosidase.

Based on the foregoing, the group research has design a randomized, double-blind, placebo-controlled crossover nutritional clinical trial to evaluate the effect of a regular probiotic with high production of beta-galactosidase effect over gastrointestinal syntoms of patients with lactose intolerance.

DETAILED DESCRIPTION:
Probiotics are defined by Food and Agriculture Organization of the United Nations and World Health Organization (FAO/WHO) as "living microorganisms that, properly administrated, confers a benefit on individual's health". Probiotics definition it's closely related to functional food concept, which encompasses either products or ingredients that are able to exert a positive impact on individual's health beyond their nutritional value. In fact, most of consumers in developed countries, strongly associate probiotics as functional foods. Lactic acid bacteria are the main microorganisms used as a probiotic, being Lactobacillus, Bifidobacterium, Propionibacterium and Streptococcus genus the most applied. Additionally, some Saccharomyces yeast may be used as probiotics.

However, a microorganism should present particular characteristic in human gastrointestinal's tract to be considered as a probiotic, following the Joint FAO/WHO Group directions: resistance to gastric and pancreatic secretions; adherence to intestinal epithelium and mucosa; antimicrobial activity against pathogenic bacteria; capability of reducing pathogen adhesion on intestinal epithelium; and present certain enzyme activity. The former bacteria genus fulfill most of the previous characteristics. However, these microorganism survival on gut is quite low (1-15%). For this reason, recent Works are searching for microorganism genus able to survive in a larger extend in gut.

Non-pathogenic bacteria of Bacillus genus have spore forming ability in the gastrointestinal tract. Specifically, Bacillus coagulans strain has been subject of new studies. B. coagulans has an optimal growth temperature of 35-50ºC, with pH conditions nearby 6. This microorganism consumes glucose, sucrose, maltose and mannitol while growing to produce lactic acid. In addition, B.coagulans is able to produce some enzymes (depending on the strain) such as alpha and beta-galactosidase, alpha-amylase, lipase and protease. However, the capability of growing in gut depends on time from its consumption (mostly oral) and the spore generation rate. The optimal dose is about 9,52x10e11 UFC, if an standard adult of 70 Kg is assumed. In addition, several studies have proved the B.coagulans ability of forming spores in presence of energy sources such as fructose and lactose.

Lactose intolerance is a chronic disease caused by the total/partial lack of lactase production. When lactose is not properly digest, it is consumed by the microbiota. This situation presents different gastrointestinal symptoms such as meteorism, pain, bloating, diarrhoea and nausea. The dietetic treatment for this patients consists of avoiding lactose-rich foods, mainly milk and dairy products. However, nowadays exists a large diversity of lactose-free products specially focused on lactose intolerants. In this context, using B.coagulans as a probiotic in a food matrix could be an alternative for these patients, since its ability of spore forming and the production of beta-galactosidase.

Based on the foregoing, the group research has designed a randomized, double-blind, placebo-controlled crossover nutritional clinical trial to evaluate the effect of a regular probiotic with high production of beta-galactosidase effect over gastrointestinal syntoms of patients with lactose intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at 18-65 years of age
* Body Mass Index (BMI) ≥18,5 and <35 kg/m2
* Patients with lactose intolerance
* Patients with a social environment that do not prevent the clinical trial fulfillment
* Patients with proper cultural level and good understanding level about the clinical trial
* Patients that have voluntarily agreed to participate in the clinical trial, giving the written informed consent.

Exclusion Criteria:

* Patients with Body Mass Index (BMI) <18,5 or ≥35 kg/m2
* Patients with Diabetes Mellitus type 1 (DMI) or Diabetes Mellitus type 2 (DMII) with no treatment
* Patients diagnosed with metabolic syndrome
* Patients diagnosed with hyperthyroidism/hypothyroidism with no treatment
* Patients with eating disorders
* Patients with diagnosed mental disorder (dementia, any cognitive function decline)
* Patients with celiac disease
* Patients with uncontrolled high blood pressure (last 2 months)
* Patients with serious disease (ascites, cirrhosis, kidney failure, heart failure, pseudomembranous colitis, lung failure, cancer, etc.)
* Patients with chronic inflammatory bowel disease (gastritis, ulcerative colitis, irritable bowel syndrome, Crohn disease, bowel perforation, etc.)
* Patients with glomerular filtration rate <90 ml/min/1,73 m2
* Patients with auto-immune diseases
* Patients undergoing corticosteroids or immunosuppressive treatment (last 12 months)
* Patients with recent episodes of nausea, vomits or diarrhoea (last 2 weeks)
* Patients with major surgery (last 3 months)
* Patients with gastrointestinal surgery (last 6 months)
* Patients with surgery for weight loss (gastric bypass, lap band)
* Patients on anticoagulation therapy
* Patients with diagnosed lactase congenital deficit
* Patients with fructose intolerance
* Patients with allergies to cow's milk protein
* Patients with intolerance to any of the ingredients of the clinical trial products.
* Patients with excessive exercise (>2h, thrice per week)
* Patients undergoing antibiotic treatment (last month)
* Patients with high consume of supplements (antioxidants, omega-3, vitamins, minerals, prebiotics) (last 2 weeks)
* Patients with regular consumption of fermented foods (≥3 times per week, such as yogurt, kefir, blue cheese) or probiotics.
* Patients with alcoholic consumptions > 30 g/d (i.e. 300 mL of wine, 3 bottles of beer, a cup of whiskey (75 mL) or similar distilled alcoholic beverages)
* Patients with regular use of laxatives (>2 per week)
* Patients participating in more clinical trials at the same time.
* Pregnant/breastfeeding women
* Women with regular use of contraception treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | 3 months
  The questionnaire developed by Casellas et al. 2009 on the specific symptoms of lactose intolerance. The patient will indicate on a scale of 1 to 10 the intensity of the following gastrointestinal symptoms: abdominal pain, bloating, flatulence, diarrhea and cramps. The scale indicates the total absence of symptoms (0) or their severe presence (10).

SECONDARY OUTCOMES:
Sensory perception | 3 months
  It is evaluated using a visual analog scale (VAS) on different sensory aspects of the product: the desire to take it, taste, smell, consistency and effectiveness of its consumption. The scale analyzes values between 0% (most negative values) or 100% (extremely positive values).
Physical activity | 3 months
  Use of International Physical Activity Questionnaire (IPAQ) to determine changes on physical activity during the clinical trial
Waist circumference | 3 months
  Data referring to the waist circumference of the Spanish population allow to estimate cardiovascular risk parameters from 95 cm in men and 82 cm in women, and very high risk from 102 cm in men and 90 cm in women. The measurement is taken at the narrowest point between the last rib and the iliac crest, with the tape against the skin but not compressed. The person should be kept in an upright position, distributing the weight equally on both legs and their arms relaxed at the sides of the body.
Body weight | 3 months
  Body weight is measured using a digital scale for clinical use (capacity 0 - 150 kg), with the person positioned with their back to the viewer, without shoes, with a minimum of warm clothing (pants and t-shirt), heels together, looking towards straight forehead and body posture.
Digestive Symptoms Questionnaire (GSRS) | 3 months
  Assessment of digestive symptoms throughout the study. The questionnaire includes 15 items grouped into 5 blocks based on different gastrointestinal symptoms. The 5 groups of symptoms are: reflux, abdominal pain, indigestion, diarrhea and constipation. Subject is asked about pain or discomfort in the upper abdomen or pit of the stomach, heartburn, acid reflux, hunger, nausea, "gut rumbling," bloating, belching, farting, constipation , diarrhoea, loose or hard stools, an urgent need to have a bowel movement and a feeling of not having finished having a bowel movement. It is scored based on a 7-point Likert-type scale, where 1 represents the most positive option and 7 the most negative. The equivalence in this questionnaire would be: 1 asymptomatic; 2 slight discomfort; 3 mild symptoms; 4 moderate symptoms; 5 moderately severe symptoms; 6 severe symptoms; 7 very serious symptoms
Changes in stool quality | 3 months
  Bristol scale to find out changes in stool form and stool frequency. The Bristol scale has 7 groups: types 1 and 2 are indicative of constipation, types 3 and 4 are desirable stools, especially 4, since they are the easiest to defecate, finally types 5, 6 and 7 are indicative diarrhea or cholera

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No